CLINICAL TRIAL: NCT07321340
Title: Insole Optimization for Rheumatoid Arthritis Patients - INORA - (Insole Optimization for Rheumatoid Arthritis Patients)
Brief Title: Insole Optimization for Rheumatoid Arthritis Patients
Acronym: INORA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: SAINBIOSE (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 25CH256; ANSM (Other: 2025-A02220-49)
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Rhumatoid Arthisis
Keywords: Insole; Rheumatoid arthritis; Feet
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D imaging (foot CT scan) (Other): foot CT scan
  Interventions: Other: gait analysis from 3D imaging (ENSENSO)

INTERVENTIONS:
Other: gait analysis from 3D imaging (ENSENSO) — gait analysis from 3D imaging (ENSENSO) on patients with bone geomtry 3D imaging

SUMMARY:
Rheumatoid arthritis affects 0.5% of the population, often leading to foot deformities and pain that are difficult to treat. Management is based on controlling inflammation, adapting footwear and using custom-made insoles, all of which have proven effective. The aim of this research is to build a digital model of plantar pressures based on CT scans, in order to optimize orthopedic insoles. The study will analyze the gait of patients with and without standard insoles to identify mechanical criteria correlated with pain. The ultimate aim is to design optimized insoles, validated by a new gait analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rheumatoid arthritis according to 2010 ACR/EULAR criteria
* RA at low activity level according to DAS28≤3.2
* Patient with mechanical forefoot involvement on walking and improved by foot orthoses.

Exclusion Criteria:

* Patients with a contraindication to a bone scan
* Patients with neurological gait disorders that interfere with gait analysis
* Exclude particularly protected persons:

  * Pregnant women, parturients, nursing mothers;
  * Persons deprived of liberty, hospitalized without consent, hospitalized for purposes other than research;
  * Minors;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Construction of a patient-specific 3D model reproducing a gait cycle with or without an orthosis. | Week 1
  Bone geometry from 3D imaging (foot CT) combined with gait analysis (speed, step length, angular variation at the knee and ankle) from 3D imaging (ENSENSO) and accelerometers

SECONDARY OUTCOMES:
Correlation of model parameters with pain | Day 1
  - Visual analogue scale (VAS) for pain in the right and left foot (0 = no pain; 10 = worst imaginable pain).
Correlation of model parameters with insole-wearing comfort. | Day 1
  Visual analogue scale (VAS) for comfort in the right and left foot (0 = most comfortable; 10 = most uncomfortable).

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Saint-Etienne, Saint-Etienne, France